CLINICAL TRIAL: NCT05370378
Title: Comparative Effects of Hold Relax With Agonist Contraction and Active Release Therapy on Pain, Functional Disability and Sleep Quality in Piriformis Syndrome
Brief Title: Effects of Hold Relax With Agonist Contraction and Active Release Therapy on Clinical Outcomes in Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Dr. Ayesha Jamil, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nimra Ilyas
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Piriformis Syndrome
Keywords: Function, Pain,Hold Relax ,Sleep Quality, Mobilization
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Group A: Hold Relax with Agonist Contraction with Routine Physical Therapy Group B: Active Release Therapy with Routine Physical Therapy
Who Masked: Outcomes Assessor
Masking Description: Opaque Sealed Envelops will be provided to participants by investigator, with mentioned treatment group. A separate therapist serving as outcome assessor will be unaware of treatment group provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group of participants will receive Hold Relax with Agonist Contraction (HR-AC) technique with routine physical therapy. The protocol will be given to the participants for two weeks (6 sessions on alternate days, 3 session per week). Each session will be of 60 minutes. The data will be collected before applying intervention, at first week and at 2nd week.
  Interventions: Other: Hold Relax with Agonist Contraction
- Group B (Active Comparator): This group of participants will receive Active Release Therapy, a kind of soft tissue mobilization along with routine physical therapy. The protocol will be given to the participants for two weeks (6 sessions on alternate days, 3 session per week). Each session will be of 60 minutes. The data will be collected before applying intervention, at first week and at 2nd week.
  Interventions: Other: Active Release Therapy

INTERVENTIONS:
Other: Hold Relax with Agonist Contraction — 1. Participant will be in prone lying and heating pad will be applied on gluteal region for 10 to 15 minutes.
  2. Passive sustained stretch to piriformis will be applied for 10 seconds.
  3. The participant will be asked to actively contract the muscle for about 10 seconds (isometric contraction) and then relax.
  4. Immediately after that participant is ask to again actively contract the muscle against therapist resistance for 6-10 seconds.
  5. Ask the participant to relax while therapist will apply stretch the muscle to its new tissue tension barrier position and this position will be maintained for 30 seconds.
  6. This maneuver is repeated for 3 to 4 repetitions, each starting from where the previous finished.
  Other Names: Proprioceptive Neuromuscular Facilitation Technique
  Arms: Group A
Other: Active Release Therapy — 1. Specific muscle will be warmed up by applying heating pad for 10 to 15 minutes.
  2. Patient will be positioned prone lying and the therapist will be standing at the side of affected limb.
  3. Therapist will apply deep pressure at the area of tenderness while patient will actively move the limb from internal to external rotation repeatedly.
  4. This maneuver will take about 15 minutes to complete in one session and will be applied alternatively 3 days a week for two weeks.
  5. After this, cold pack is applied and general ROMs and strengthening exercises are performed to prevent soreness
  Other Names: Soft Tissue Mobilization
  Arms: Group B

SUMMARY:
The aim of this study is to compare the effects of hold relax agonist contraction and active release therapy on reducing pain intensity, improving functioning and sleep quality in patient with piriformis syndrome.

Both these techniques are passive, non-invasive manual therapy techniques which are easy to perform and less time consuming and may yield better outcomes resulting improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 25-55 years
2. Both male and female.
3. Gluteal pain with or without radicular symptoms.
4. Patients of piriformis syndrome diagnosed by orthopedic consultant.
5. Sub-acute and chronic piriformis syndrome.
6. Unilateral pain.
7. Pain score equal to and greater than 3 according to pain rating scale.

Exclusion Criteria:

1. Intermittent vascular claudication and spondylolisthesis.
2. Past history of hip, femur or vertebral fracture
3. Past history of spinal surgery.
4. Spinal tuberculosis.
5. Rheumatoid disease.
6. Disc pathology, sacroiliac joint dysfunction or mechanical back pain.
7. History of infectious disease.
8. Leg length discrepancy.
9. Any postural abnormality or deformity.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | Pain score will be measured at the baseline, at end of first session and at 6th session on 2nd week
  Numeric Pain Rating Scale will be used to measure the intensity of pain
Change in Functional Disability | Change in functional status will be measured at the baseline, at end of first session and at end of 6th session
  Ronald-Morris Disability Questionnaire will be used to a assess the level of disability
Sleep Quality | Sleep quality will be measured at the baseline, at end of first session and at end of 6th session
  Chronic Pain Sleep Inventory will be used to to assess the quality of sleep on a 100 mm VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Jamil, M.Phil, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies the results reported in article after deidentification
Supporting Information: Study Protocol
Time Frame: Immediately following publication. Ending in 36 months.